CLINICAL TRIAL: NCT06361342
Title: Smartphones Aggravating Anxiety Symptoms: Experimental Study From Southeastern
Brief Title: Smartphones Aggravating Anxiety Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gagandeep Singh, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-003633
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anxiety
Keywords: Smartphones
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General decrease in smartphone use. (Experimental): Subjects will limit their time on smartphone.
  Interventions: Behavioral: General decrease in smartphone use
- Avoid certain social media apps (Experimental): Subjects will limit time on smartphone, in particular avoiding use of social media apps on the smartphone which includes Twitter, Facebook, Tik Tok, Instagram, and Pinterest.
  Interventions: Behavioral: Avoiding Social Media Apps

INTERVENTIONS:
Behavioral: General decrease in smartphone use — Subjects will decrease their time on smartphone in general.
  Arms: General decrease in smartphone use.
Behavioral: Avoiding Social Media Apps — Subjects will avoid use of social media apps on the smartphone which includes Twitter, Facebook, Tik Tok, Instagram, and Pinterest.
  Arms: Avoid certain social media apps

SUMMARY:
The goal of this study is to assess if excessive use of smartphone apps of social media can impact a person's mental health. The study is aimed at improving the usage of smartphones which might help improve the mental health of patients. The goal is not to discourage the use of smartphones but instead to utilize smartphones in a way that they do not impact lives.

ELIGIBILITY:
Inclusion Criteria:

* For patients aged 18 years or older experiencing mild symptoms of anxiety or depression and who have a GAD-7 score 5 and above.
* Patient should have smart phone and should be using Facebook, Instagram, Twitter, Tik Tok, and Pinterest social media apps.
* Patients should have email access.

Exclusion Criteria:

* Any patient who uses a smartphone for tracking glucose for diabetes management, heart rate, or any chronic illness which is being managed through a smartphone app.
* Any patient who uses more than one personal smartphone
* Any patient who is a suicide risk as per PHQ-9 score, current recreational drug usage, or alcohol abuse.
* Any patient who has suicidal ideation as per PHQ-9 assessment before or during the study period will be excluded, (all patients will be monitored for suicidal ideation by PHQ-9 scoring method at day 1, week 6, and week 12, but it is the responsibility of the patient to inform the study team if they have developed any suicidal ideation throughout the study period).
* Patients with activated POA (Power of Attorney - Healthcare), diagnosis of mental retardation or current disability due to any psychiatric disorder or severe depression with a high risk of suicide should be excluded.
* Any patient currently undergoing ECT (electroconvulsive therapy) for severe depression.
* Any patient taking prescribed SSRIs/SNRIs, with a change and not taking them continuously in last 30 days (not a new diagnosis of anxiety). If change they will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety | Day 1, 12 weeks
  Measured using the General Anxiety Disorder 7-item (GAD 7) scale to assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety.

SECONDARY OUTCOMES:
Change in depression | Day 1, 12 weeks
  Measured using the Patient Health Questionnaire 9-item (PHQ-9) scale used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Gagandeep Singh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No